CLINICAL TRIAL: NCT03758118
Title: Neuroprotection and Neuroenhancement in a Model of Optic Nerve Neurodegeneration (Non Arteritic Ischemic Optic Neuropathy): Study of Morpho-functional Changes Related to Treatment With Citicoline Oral Solution
Brief Title: Citicoline in Non-Arteritic Ischemic Optic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione G.B. Bietti, IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 85356727
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Results first posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2021-02

CONDITIONS: Non-arteritic Ischemic Optic Neuropathy
Keywords: Citicoline; Non-arteritic ischemic optic neuropathy; Neuroprotection; Neuroenhancement
MeSH Terms: interventions — Cytidine Diphosphate Choline

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAION patients OS-Citicoline treated (Active Comparator): In a group of patients with NAION, OS-Citicoline will be administered (500 mg/day) for 6 months followed by three months of suspension
  Interventions: Dietary Supplement: Citicoline
- NAION patients untreated (No Intervention): In one group of patients with NAION no type of treatment will be performed during 9 months of observation

INTERVENTIONS:
Dietary Supplement: Citicoline — Citicoline administered in oral solution
  Arms: NAION patients OS-Citicoline treated

SUMMARY:
The investigators tested the hypothesis whether the treatment with Citicoline in oral solution (OS-Citicoline) would increase or stabilize visual acuity, retinal ganglion cells (RGCs) function and neural conduction along the visual pathways (neuroenhancement), and/or induce preservation of RGCs fibers' loss (neuroprotection) in an human model of neurodegeneration: non-arteritic ischemic optic neuropathy (NAION).

DETAILED DESCRIPTION:
The investigators enrolled 40 patients with bilateral or monolateral NAION and 20 age similar controls

Twenty NAION patients received 500 mg/day of OS-Citicoline for a 6-months period followed by 3-months of wash-out (19 patients completed the study, NC Group); 20 NAION patients were not treated (19 patients completed the studyNN Group) from baseline up to 9 months. In all subjects, at baseline, at 6 and 9-months of follow-up: Visual acuity (VA), Pattern Electroretinogram (PERG), Visual Evoked Potentials (VEP), retinal nerve fiber layer thickness (RNFL-T) and Humphrey 24-2 visual field mean deviation (HFA MD) were assessed. Mean differences were statistically evaluated by ANOVA between Groups, and correlations were verified by Pearson's test.

ELIGIBILITY:
Inclusion criteria:

1. Acute visual reduction episode from NAION occurring for more than 6 months
2. Typical defects of the visual field evidenced with the Goldmann perimetry or with Humphrey perimetry 30-2
3. Visual acuity not less than 1/10
4. Having suspended any potential neuroprotective therapies (e.g., Coenzyme Q10) for at least 6 months.

Exclusion criteria:

* Ocular surgery in the 3 months preceding the study, including surgery for cataracts in the previous three months.
* Cataract or maculopathy
* Known hypersensitivity to the study product
* Positive history for diseases of the optic nerve (retrobulbar optic neuropathy, glaucoma) or systemic diseases which could preclude the enrolment in the study according to the investigators' judgement
* Pregnant or nursing women, or women of potential childbearing age not using adequate contraception.
* Diabetes, SLE, rheumatoid arthritis, mixed connective tissue disease

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2017-07-25 (Actual); Study Completion 2018-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo MF Parisi, MD, Principal Investigator — Fondazione Bietti- IRCCS
Locations (1):
- Britannico Hospital, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carelli V, La Morgia C, Ross-Cisneros FN, Sadun AA. Optic neuropathies: the tip of the neurodegeneration iceberg. Hum Mol Genet. 2017 Oct 1;26(R2):R139-R150. doi: 10.1093/hmg/ddx273. PMID 28977448
- [Background] Cho YS. The role of necroptosis in the treatment of diseases. BMB Rep. 2018 May;51(5):219-224. doi: 10.5483/bmbrep.2018.51.5.074. PMID 29636122
- [Background] Hayreh SS, Zimmerman B. Visual field abnormalities in nonarteritic anterior ischemic optic neuropathy: their pattern and prevalence at initial examination. Arch Ophthalmol. 2005 Nov;123(11):1554-62. doi: 10.1001/archopht.123.11.1554. PMID 16286618
- [Background] Patel HR, Margo CE. Pathology of Ischemic Optic Neuropathy. Arch Pathol Lab Med. 2017 Jan;141(1):162-166. doi: 10.5858/arpa.2016-0027-RS. PMID 28029908
- [Background] Parisi V, Gallinaro G, Ziccardi L, Coppola G. Electrophysiological assessment of visual function in patients with non-arteritic ischaemic optic neuropathy. Eur J Neurol. 2008 Aug;15(8):839-45. doi: 10.1111/j.1468-1331.2008.02200.x. Epub 2008 Jun 28. PMID 18557920
- [Background] Balducci N, Morara M, Veronese C, Barboni P, Casadei NL, Savini G, Parisi V, Sadun AA, Ciardella A. Optical coherence tomography angiography in acute arteritic and non-arteritic anterior ischemic optic neuropathy. Graefes Arch Clin Exp Ophthalmol. 2017 Nov;255(11):2255-2261. doi: 10.1007/s00417-017-3774-y. Epub 2017 Aug 31. PMID 28861697
- [Background] Khalilpour S, Latifi S, Behnammanesh G, Majid AMSA, Majid ASA, Tamayol A. Ischemic optic neuropathy as a model of neurodegenerative disorder: A review of pathogenic mechanism of axonal degeneration and the role of neuroprotection. J Neurol Sci. 2017 Apr 15;375:430-441. doi: 10.1016/j.jns.2016.12.044. Epub 2016 Dec 26. PMID 28320183
- [Derived] Parisi V, Barbano L, Di Renzo A, Coppola G, Ziccardi L. Neuroenhancement and neuroprotection by oral solution citicoline in non-arteritic ischemic optic neuropathy as a model of neurodegeneration: A randomized pilot study. PLoS One. 2019 Jul 26;14(7):e0220435. doi: 10.1371/journal.pone.0220435. eCollection 2019. PMID 31348806

RESULTS

PARTICIPANT FLOW:
Groups:
- NAION Patients OS-Citicoline Treated: In 20 patients with NAION, OS-Citicoline was administered (500 mg/day) for 6 months followed by three months of suspension (19 completed the study, NC Group)
  Citicoline: Citicoline administered in oral solution
- NAION Patients Untreated: In 20 patients with NAION no type of treatment was performed during 9 months of observation (17 patients completed the study, NN Group)
Period: Overall Study
Arm/Group | NAION Patients OS-Citicoline Treated | NAION Patients Untreated
Started | 20 | 20
Completed | 19 | 17
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Units Other Than Participants: eyes
Groups:
- NAION Patients OS-Citicoline Treated: In 20 patients with NAION, OS-Citicoline will be administered (500 mg/day) for 6 months followed by three months of suspension (NC Group)
- NAION Patients Untreated: In 20 patients with NAION, no type of treatment will be performed during 9 months of observation (NN Group)
- Total: Total of all reporting groups
Arm/Group | NAION Patients OS-Citicoline Treated | NAION Patients Untreated | Total
Number analyzed (Participants) | 20 | 20 | 40
Number analyzed (eyes) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 23
  >=65 years | 9 | 8 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 20 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 20 | 20 | 40
Number of Participants with NAION diagnosis in the last 6 - 12 months [Count of Participants; unit: Participants] | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Visual Acuity at 9 Month
Description: Increase of Visual Acuity evaluated by Early Treatment Diabetic Retinopathy Study (ETDRS) charts and measured as a logarithm of the minimum angle of resolution (LogMAR)
Time Frame: 9 months vs baseline
Measure: Mean (Standard Deviation); unit: LogMAR
Groups:
- NAION Patients OS-Citicoline Treated: 19 eyes completed the study, 1 eye drop-out
- NAION Patients Untreated: 17 eyes completed the study, 3 eyes drop-out
Arm/Group | NAION Patients OS-Citicoline Treated | NAION Patients Untreated
Number analyzed (Participants) | 19 | 17
LogMAR | -0.0574 (0.1147) | 0.0535 (0.0914)

2. Secondary Outcome: Change From Baseline in Retinal Ganglion Cells Function at 9 Month
Description: Pattern-Electroretinogram recordings. Increase of P50-N95 amplitude (measured in microvolt)
Time Frame: 9 months vs Baseline
Measure: Mean (Standard Deviation); unit: microvolt
Arm/Group | NAION Patients OS-Citicoline Treated | NAION Patients Untreated
Number analyzed (Participants) | 19 | 17
microvolt | 1.32 (0.39) | 1.38 (0.28)

3. Secondary Outcome: Change From Baseline in Optic Nerve Function at 9 Months
Description: Visual Evoked Potentials recordings. Shortening of the main parameter P100 Implicit time measured in milliseconds
Time Frame: 9 months vs baseline
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | NAION Patients OS-Citicoline Treated | NAION Patients Untreated
Number analyzed (Participants) | 19 | 17
milliseconds | 127.05 (8.35) | 126.88 (6.50)

4. Secondary Outcome: Change From Baseline in Optic Nerve Morphology at 9 Months
Description: Reduction of Overall Retinal Nerve Fiber Thickness by Optical Coherence Tomography measured in micron
Time Frame: 9 months vs baseline
Measure: Mean (Standard Deviation); unit: micron
Arm/Group | NAION Patients OS-Citicoline Treated | NAION Patients Untreated
Number analyzed (Participants) | 19 | 17
micron | 57.71 (9.43) | 63.99 (8.44)

5. Secondary Outcome: Change From Baseline in Visual Field Defects at 9 Months
Description: improvement of the visual field by static perimetry (increase of the main indexes Mean Deviation measured in dB).
Time Frame: 9 months vs baseline
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | NAION Patients OS-Citicoline Treated | NAION Patients Untreated
Number analyzed (Participants) | 19 | 17
dB | -15.61 (6.43) | -13.02 (7.15)

ADVERSE EVENTS:
Time Frame: 9 months
Description: No adverse events were observed in any patient enrolled
Groups:
- NAION Patients OS-Citicoline Treated: 19 NAION patients providing 19 eyes completed the study
- NAION Patients Untreated: 17 NAION patients providing 17 eyes completed the study
Arm/Group | NAION Patients OS-Citicoline Treated | NAION Patients Untreated
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/17
Other Adverse Events (participants affected / at risk) | 0/19 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-20): https://cdn.clinicaltrials.gov/large-docs/18/NCT03758118/Prot_SAP_000.pdf